CLINICAL TRIAL: NCT03364478
Title: Randomized Controlled Trial: Comparative Study of Medial-to-Lateral Approach vs Dorsal and Medial Hybrid Approach in Laparoscopic Right Hemicolectomy
Brief Title: Comparative Study of Medial-to-Lateral Approach vs Dorsal and Medial Hybrid Approach in Laparoscopic Right Hemicolectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ShanghaiMISC-RHC
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Overall Survival; Postoperative Complications
Keywords: Surgical approach; Laparoscopic right hemicolectomy
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DML group (Experimental): The group underwent laparoscopic right hemicolectomy with dorsal and medial hybrid approach. In DML group, the dissecting based on CME is performed with dorsal approach and medial approach hybridized.
  Interventions: Procedure: DML group
- MLA group (Active Comparator): The group underwent laparoscopic right hemicolectomy with traditional medial-to-lateral approach. In MLA group,the dissecting based on CME is performed with meidial-to-lateral approach.
  Interventions: Procedure: MLA group

INTERVENTIONS:
Procedure: DML group — The group underwent laparoscopic right hemicolectomy with dorsal and medial hybrid approach.
  Arms: DML group
Procedure: MLA group — The group underwent laparoscopic right hemicolectomy with traditional medial-to-lateral approach.
  Arms: MLA group

SUMMARY:
To standardize the surgery for advanced right hemi colon cancer with laparoscopy and investigate whether dorsal and medial hybrid approach could improve disease-free survival in patients with right colon cancer, compared with traditional medial-to-lateral approach in laparoscopic righ hemicolectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged more then 18 years old;
* Diagnosed as right hemi colonic cancer with colonoscopic biopsy;
* Without metastasis;
* No Invasion of surrounding tissues;
* Limited operation;
* Underwent laparoscopic radical right hemicolectomy (L-right hemicolectomy);
* BMI 18~30kg/m2;
* Without multiple primary tumors;
* Sign on the Medical informed Consent.

Exclusion Criteria:

* Simultaneous or simultaneous multiple primary colorectal cancer;
* Preoperative imaging examination results show:

  1. Tumor involves the surrounding organs and combined organ resection need to be done;
  2. Distant metastasis;
  3. Unable to perform R0 resection;
* History of any other malignant tumor in recent 5 years;
* Patients need emergency operation;
* Not suitable for laparoscopic surgery;
* Women during Pregnancy or breast feeding period;
* Informed consent refusal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
The rate of postoperative complication | 30 days
3 years overall survival | 3 years
The rate of local and distant recurrence | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, PhD, Study Director — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospttal, Shanghai, Sahgnhai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fujita J, Uyama I, Sugioka A, Komori Y, Matsui H, Hasumi A. Laparoscopic right hemicolectomy with radical lymph node dissection using the no-touch isolation technique for advanced colon cancer. Surg Today. 2001;31(1):93-6. doi: 10.1007/s005950170230. PMID 11213054
- [Result] Matsuda T, Iwasaki T, Mitsutsuji M, Hirata K, Maekawa Y, Tanaka T, Shimada E, Kakeji Y. Cranial-to-caudal approach for radical lymph node dissection along the surgical trunk in laparoscopic right hemicolectomy. Surg Endosc. 2015 Apr;29(4):1001. doi: 10.1007/s00464-014-3761-x. Epub 2014 Aug 19. PMID 25135445
- [Result] Li H, He Y, Lin Z, Xiong W, Diao D, Wang W, Wan J, Zou L. Laparoscopic caudal-to-cranial approach for radical lymph node dissection in right hemicolectomy. Langenbecks Arch Surg. 2016 Aug;401(5):741-6. doi: 10.1007/s00423-016-1465-5. Epub 2016 Jun 18. PMID 27318491
- [Result] Zou L, Xiong W, Mo D, He Y, Li H, Tan P, Wang W, Wan J. Laparoscopic Radical Extended Right Hemicolectomy Using a Caudal-to-Cranial Approach. Ann Surg Oncol. 2016 Aug;23(8):2562-3. doi: 10.1245/s10434-016-5215-2. Epub 2016 Apr 12. PMID 27072997
- [Result] Lotti M, Capponi MG, Campanati L, Bertoli P, Palamara F, Coccolini F, Ansaloni L. Laparoscopic right colectomy: Miles away or just around the corner? J Minim Access Surg. 2016 Jan-Mar;12(1):41-6. doi: 10.4103/0972-9941.158960. PMID 26917918
- [Result] Zheng B, Wang N, Wu T, Qiao Q, Zhou S, Zhang B, Yang Y, Xie S, Wang K, He X. [Comparison of cranial-to-caudal medial versus traditional medial approach in laparoscopic right hemicolectomy: a case-control study]. Zhonghua Wei Chang Wai Ke Za Zhi. 2015 Aug;18(8):812-6. Chinese. PMID 26303693
- [Result] Honaker M, Scouten S, Sacksner J, Ziegler M, Wasvary H. A medial to lateral approach offers a superior lymph node harvest for laparoscopic right colectomy. Int J Colorectal Dis. 2016 Mar;31(3):631-4. doi: 10.1007/s00384-015-2499-9. Epub 2016 Jan 22. PMID 26801787